CLINICAL TRIAL: NCT03659097
Title: Evaluation of the Efficacy of Periodontally Accelerated Osteogenic Orthodontics in the Leveling and Alignment of Crowded Lower Anterior Teeth: A Two-Arm Randomized Controlled Clinical Trial
Brief Title: Acceleration of Alignment of Crowded Lower Anterior Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-17-2018
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Malocclusion, Angle Class I; Crowded Teeth
MeSH Terms: conditions — Malocclusion, Angle Class I; Crowding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontally accelerated osteogenic orthodontics (Experimental): Patients in this group will undergo orthodontic treatment plus periodontally accelerated osteogenic orthodontics in order to induce tooth movement.
  Interventions: Procedure: periodontally accelerated osteogenic orthodontics
- Traditional orthodontics (No Intervention): Patients in this group will undergo traditional orthodontics without any surgical interventions

INTERVENTIONS:
Procedure: periodontally accelerated osteogenic orthodontics — Surgery will be performed to the lower anterior bony segment of the lower jaw in order to accelerate tooth movement
  Other Names: PAOO
  Arms: Periodontally accelerated osteogenic orthodontics

SUMMARY:
Patients at the Orthodontic Department of University of Damascus Dental School will be examined and subjects who meet the inclusion criteria will be included. Then, initial diagnostic records (diagnostic gypsum models, internal and external oral photographs, as well as radiographic images) will be studied to ensure that the selection criteria are accurately matched.

The aim of this study is to compare two groups of patients with moderate crowding of the lower anterior teeth First group (Experimental): the patients in this group will be treated with orthodontic fixed appliances + surgery to the alveolus of the lower anterior teeth in order to induce remodeling of the bony structures and enhance orthodontic movement.

Second group (Control): the patients in this group will be treated using fixed appliances with any acceleration method.

ELIGIBILITY:
Inclusion Criteria:

* Class I malocclusion with moderate crowding (4-6 mm of tooth-size-arch-length-discrepancy).
* Good oral hygiene and periodontal health.
* No severe skeletal discrepancy.
* Normal inclination for the upper and lower incisors.
* No congenitally missing or extracted teeth (except for the third molars).

Exclusion Criteria:

* Bi-maxillary severe dental protrusion.
* Previous orthodontic treatment.
* Subject with psychological abnormalities.
* Subject with systemic diseases.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-09-02 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Duration of Alignment | The assessment is based on calculating days from the beginning of treatment till the end of the alignment stage which is expected to happen within 5 to 6 months
  The time required in days will be calculated from the beginning of treatment till the end of the alignment stage
Change in Little's Index of Irregularity | T0: one day before the beginning of treatment; T1: after 1 month; T2: after 2 months; T3: after 4 months; T4: after 5 months; T5: at the end of the alignment stage which is expected within 5 - 6 months
  The irregularity of the lower incisors is calculated by measuring the amount of deviations of the anatomic contact points between the six anterior teeth in the horizontal direction in mm, since the sum of these measurements represents the value of the index (Little, 1975). When the sum of these deviations is less than 3 mm, this indicates that the teeth are slightly crowded. When the sum is greater than 10 mm, this indicated very severe crowding.
  The ordinary orthodontic treatment aims to keep this Index less than 1 mm at the end of treatment.
Change in Alveolar Defect | T1: One day before the beginning of treatment; T2: at the end of the alignment stage which is expected within 5-6 months
  Using cone-beam computed tomography (CBCT), each tooth root will be evaluated in axial and cross-sectional slices at the buccal and lingual surfaces. When no cortical bone is observed around the root in at least three sequential views, this will be considered an alveolar defect. If the alveolar bone height is more than 2 mm from the cemento-enamel junction, it will be classified as dehiscence ,When the defect does not involve the alveolar crest, this case will be classified as fenestration.
  The status of the alveolar bone will be assessed twice.

SECONDARY OUTCOMES:
Change in inter-canine width | T1: One day before the beginning of treatment; T2: at the end of the alignment stage which is expected within 5-6 months
  The distance between the cusp tips of the lower canines. This variable will be measured on plaster models.
  T1: One day before the beginning of treatment; T2: at the end of the alignment stage
Change in Alveolar Bone Thickness | T1: One day before the beginning of treatment; T2: at the end of the alignment stage which is expected within 5-6 months
  Will be measured for each of the lower anterior teeth in the cervical, middle, and apical regions. This will be achieved by using the ruler which will be positioned perpendicular to tooth long axis from the root surface (without measuring the periodontal ligament ) to the most external surface of the cortical bone.
Change in Lower Incisors' Inclination | T1: One day before the beginning of treatment; T2: at the end of the alignment stage which is expected within 5-6 months
  The angle between the long axis of the lower Incisors and the mandible plane (Go-Me) will be measured.
Change in the positioning of the upper lip | T1: One day before the beginning of treatment; T2: at the end of the alignment stage which is expected within 5-6 months
  It is going to be evaluated by Ricketts' analysis (E-Line). This is done by drawing a reference line between the tip of the nose and the most prominent point on the chin contour (Pogonion).
  The distance of the upper lip from this line is a measure of lip positioning.
Change in the positioning of the lower lip | T1: One day before the beginning of treatment; T2: at the end of the alignment stage which is expected within 5-6 months
  It is going to be evaluated by Ricketts' analysis (E-Line). This is done by drawing a reference line between the tip of the nose and the most prominent point on the chin contour (Pogonion).
  The distance of the lower lip from this line is a measure of lower lip positioning.
Change in the naso-labial angle | T1: One day before the beginning of treatment; T2: at the end of the alignment stage which is expected within 5-6 months
  It is the angle formed between the lower border of the nose and the upper lip.

CONTACTS AND LOCATIONS:
Overall Officials: Hallaj I Alsino, DDS, Principal Investigator — MSc student at the Orthodontic Department, University of Damascus Dental School, Damascus, Syria; Mohammad Y Hajeer, DDS MSc PhD, Study Director — Associate Professor of Orthodontics, University of Damascus Dental School, Damascus, Syria; Issam Khoury, DDS MSc PhD, Study Director — Professor of Oral and Maxillofacial Surgery, Oral and Maxillofacial Surgery Department, University of Damascus Dental School, Damascus, SYRIA
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munoz F, Jimenez C, Espinoza D, Vervelle A, Beugnet J, Haidar Z. Use of leukocyte and platelet-rich fibrin (L-PRF) in periodontally accelerated osteogenic orthodontics (PAOO): Clinical effects on edema and pain. J Clin Exp Dent. 2016 Apr 1;8(2):e119-24. doi: 10.4317/jced.52760. eCollection 2016 Apr. PMID 27034749
- [Background] Bahammam MA. Effectiveness of bovine-derived xenograft versus bioactive glass with periodontally accelerated osteogenic orthodontics in adults: a randomized, controlled clinical trial. BMC Oral Health. 2016 Nov 30;16(1):126. doi: 10.1186/s12903-016-0321-x. PMID 27903250
- [Background] Yu H, Jiao F, Wang B, Shen SG. Piezoelectric decortication applied in periodontally accelerated osteogenic orthodontics. J Craniofac Surg. 2013;24(5):1750-2. doi: 10.1097/SCS.0b013e3182902c5a. PMID 24036771
- [Background] Nowzari H, Yorita FK, Chang HC. Periodontally accelerated osteogenic orthodontics combined with autogenous bone grafting. Compend Contin Educ Dent. 2008 May;29(4):200-6; quiz 207, 218. PMID 18533317
- [Background] Amit G, Jps K, Pankaj B, Suchinder S, Parul B. Periodontally accelerated osteogenic orthodontics (PAOO) - a review. J Clin Exp Dent. 2012 Dec 1;4(5):e292-6. doi: 10.4317/jced.50822. eCollection 2012 Dec 1. PMID 24455038